

#### **PROJECT TITLE:**

# ASSESSMENT OF TEARS, CORNEAL STAINING AND COMFORT LEVEL AFTER ONE DAY WEAR OF CONTACT LENSES OF DIFFERENT FDA CATEGORIES AMONG UNDERGRADUATE STUDENTS OF UKM KUALA LUMPUR CAMPUS

#### **INVESTIGATORS:**

ASSOC PROF DR. HALIZA ABDUL MUTALIB (Chief Investigator)

DR. BASHIRAH ISHAK (Co-Investigator)

MR MOHD NORHAFIZUN MOHD SAMAN (Clinic Researcher)

MR ASYRAF ZULHAKIM BIN SHAMSUL (Site Investigator)

MS NUR NALIESYA BINTI ASHA'RI (Site Investigator)

MS NUR NATASHA SOFEA BINTI NICK HAMASHOLDIN (Site Investigator)

| CONTENT | TOPICS | Page |
|---------|----------------------------------------------|------|
| 1.0 | Research Topics | |
| 2.0 | Introduction | |
| 2.1 | Research Background | 1 |
| 2.2 | Problem Statement and Research Justification | 3 |
| 2.3 | Research Question | 3 |
| 2.4 | Hypothesis | 3 |
| 2.5 | Conceptual framework | 4 |
| 2.6 | Research Objective | 5 |
| 3.0 | Methodology | |
| 3.1.1 | Research Design | 6 |
| 3.1.2 | Sampling Methods | 6 |
| 3.1.3 | Study Location | 6 |
| 3.1.4 | Study Sample Calculation | 6 |
| 3.1.5 | Subject | 7 |
| 3.1.6 | Participation Criteria | 7 |
| 3.1.7 | Exclusion Criteria | 7 |
| 3.1.8 | Instrument | 7 |
| 3.1.9 | Study Protocol | 8 |
| 3.1.10 | Flowchart | 11 |
| 3.1.11 | Data Analysis | 12 |
| 4.0 | Ethical Approval | 12 |
| 5.0 | Gantt chart | 13 |
| 6.0 | Reference | 14 |

#### 1.0 STUDY TITLE

Assessment of Tears, Corneal Staining and Comfort Level After One Day Wear Of Contact Lenses Of Different FDA Categories Among Undergraduate Students of UKM Kuala Lumpur Campus.

#### 2.0 INTRODUCTION

2.1 The Food and Drug Administration (FDA) classifies soft contact lens materials into 5 groups, where hydrogels are in Group I, II, III, and IV, while silicone hydrogel (SH) is in Group V. Hydrogel silicone contact lenses are one of the results of contact lens innovations that were first introduced in the market in the late 90s (Sulley & Dumbleton, 2020). Silicone material allows for high oxygen permeability while hydrogel components maintain the softness and comfort of contact lenses (Gasson & Morris, 2003). The Group I FDA contact lens is a non-ionic hydrogel with the water content of <50%. Group II, on the other hand, is a non-ionic hydrogel with the water content of >50% (Peral et al. 2020). As for group III and IV contact lenses, they are ionic contact lenses. Group III contact lenses have a low water content of less than 50% compared to group IV with high water content of more than 50% (Peral et al. 2020). There are several examples of soft contact lens materials for each group, Polymacon and Crofilcon are examples of group I while Nelfilcon A and Omafilcon A are material examples of group II soft contact lenses. Examples of group III soft contact lens materials are Bufilcon A and Deltafilcon A while Ocufilcon B and Ocufilcon C are examples of group IV soft contact lens materials (Chatterjee et al. 2020). Material Lotrafilcon A and Balafilcon A are examples of group V soft contact lens material (Efron et al., 2010).

Protein deposits can result in multiple immune responses, including giant papillary conjunctivitis. Silicone hydrogel (SH) material contact lenses provide comfort and better performance compared to hydrogel material. The data show that very low protein deposits are present in silicone hydrogel material contact lenses after wear when compared with hydrogel material (Subbaraman et al., 2006). The application of contact lenses can cause changes in the level of production and tear quality. This can cause a feeling of discomfort in the eyes when wearing contact lenses (Fonn 2007; Maruyama et al., 2004). Based on the classification of dry eye diagnostics from the National Eye Institute and Industry Workshop, dry eye problems during contact lens wear are related to tear loss through evaporation (Lemp 1995; Pflugfelder et al., 2000). Studies from Asharlous et al. (2016) have also shown that there are significant

Date: 2/4/2024

changes in the quality and quantity of tears after 6 hours of wearing hydrogel silicone contact lenses of the Air Optix Aqua brand, Lotrafilcon B from CIBA Vision. The level of tear production can be measured by the Schirmer test; together or without anesthetic, in which it represents the secretion of tears on the lower part of the eyelid and tear reflexes. The Schirmer test is still used for the measurement of tear production in primary eye care as it is simple, fast, cheap and practical (Razak et al., 2018). The Non-Invasive Breakup Time (NIBUT) test allows stability and tear quality to be studied without inserting foreign material into the eye. This method is more patient-friendlier and more accurate than the Tear Breakup Time (TBUT) Test method. The TBUT method is considered to have a deficiency because the presence of sodium fluorescein alters the physiology of tears (Mohidin et al., 2002). Finally, a questionnaire will be used to study the level of comfort throughout the wearing of contact lenses using the Contact Lens Discomfort Index (CLDI) questionnaire, Cristina Arroyo-del Arroyo et al. (2022). The choice of questions in this questionnaire is based on the existing questionnaire Contact Lens Dry Eyes Questionnaire (CLDEQ)-8. CLDI is a strong and reliable questionnaire and this questionnaire is designed to measure the comfort level of contact lens wearing (Arroyo-del Arroyo et al., 2022).

Contact lenses are not only used to replace the wearing of glasses but are also used for treatments and cosmetic purposes. It is estimated that there are 140 million contact lens wearers worldwide (Cope et al. 2017). Therefore, it is not surprising that the wearing of contact lenses is the latest follow-up. However, contact lens wearers need to know which type of contact lenses are suitable for everyday activities. This is because, as soon as the contact lenses are placed on the eye, the lens will be on the tear film.

The ability of a tear film to maintain its integrity in the presence of lenses is a prerequisite basis for the successful application of contact lenses. Lack of interaction between tears and lenses is the most common reason for contact lens wear failure (Downie & Craig., 2017). The most common symptoms reported by contact lens wearers are dryness and discomfort in the eyes (Nursyuhada. 2021).

Date: 2/4/2024

2.1 LITERATURE REVIEW

Contact lens materials are classified by the Food and Drug Administration (FDA) and international organizations based on water content and balanced ionic properties, aligning with

their clinical performance impact. Group I lenses, with low water content and non-ionic

properties, tend to be the most stable and least influenced by tear film and environmental factors.

Conversely, Group IV lenses, characterized by high water content and ionic properties, are more

reactive and prone to interaction with positively charged proteins like lysozyme, with potential

impacts from different pH solutions. Group II and III lenses fall between these extremes and

exhibit varying performances (Jones & Dumbleton, 2019).

Over recent decades, the evolution of contact lens materials to meet consumer demands has

posed a significant challenge for manufacturers. Consequently, numerous studies have been

undertaken to evaluate ocular comfort levels associated with various types of contact lenses,

such as hydrogel and hydrogel silicone lenses. Mutalib et al. (2018) demonstrated no significant

difference in comfort levels between female students at Universiti Kebangsaan Malaysia KL

Campus when wearing hydrogel versus silicone hydrogel lenses.

Assessment of contact lens application typically occurs before and after lens wear. Ocular

comfort during lens wear depends on the interaction between the lens and ocular tissue, the

wearer's ocular physiological state, and their adherence to lens wear. Mutalib et al. (2018)

highlighted the significant impact of mechanical interaction between lens and ocular surfaces

on comfort levels. Additionally, a study by Santodomingo, Rubito et al. (2010) found no

significant difference in comfort levels between hydrogel and hydrogel silicone lenses, with

both showing a decrease in comfort after a day of wear.

Conventional hydrogel lenses often feature high water content to enhance oxygen permeability,

yet this can lead to increased dehydration and potential physiological eye disorders (Ruiz-

Alcocer et al., 2018). Ruiz-Alcocer et al. (2018) demonstrated that disposable contact lenses

can mitigate some issues associated with prolonged wear. Efforts to improve conventional

lenses include the introduction of new hydrogels with a water content of 78%. Furthermore,

5

Date: 2/4/2024

studies by Ruiz-Alcocer et al. (2018) found no difference in tear osmolality between contact lenses, suggesting that tear dryness symptoms may not be significantly impacted by lens type.

The corneal epithelium and conjunctiva play crucial roles in protecting the cornea and conjunctival layers. It's widely acknowledged that epithelial disorders can predispose individuals to fungal, viral, or bacterial eye infections. However, research also indicates that corneal infections can stem from conditions involving cellular epithelium, tear film biochemistry, and bacterial resistance to epithelial basal lamina (Brautaset et al., 2008).

In wearers of hydrogel soft contact lenses, staining on the conjunctival epithelium may result from various physical factors such as pressure from the lens edge, edge defects, and lens removal techniques (Brautaset et al., 2008).

Lakkis and Brennan (1996) conducted a study involving 50 hydrogel contact lens wearers and 50 non-contact lens wearers, revealing that 98% of lens wearers exhibited some degree of corneal staining compared to only 12% of non-wearers. Moreover, 62% of lens wearers experienced corneal staining exceeding grade 1 on the Efron scale.

Corneal staining in hydrogel contact lens wearers is attributed to tear film dysfunction, hypoxia, mechanical forces, exposure, metabolic disorders, toxic or allergic reactions, and infectious reactions. The prevalence of corneal staining in hydrogel contact lens wearers ranges from approximately 30% to 55.7% (Brautaset et al., 2008). Nicholas et al. (2000) also noted associations between staining presence and levels with non-compliance regarding contact lens care systems, use of rewetting drops, and absence of a lens replacement plan. However, no associations were found with age, gender, medications, continued wear versus daily wear, wearing time, lens type, water content, or contact lens care system (Brautaset et al., 2008).

Research by Nicholas and Sinnott (2006) revealed a higher likelihood of dry eyes associated with the use of high water content contact lenses. However, lens ionization was not found to be linked to dry eye symptoms. In a subsequent analysis, they demonstrated that compared to Group I FDA contact lenses, both Group II and IV FDA lenses were associated with a 2-3 times increase in the likelihood of dry eyes for contact lens wearers. Additionally, in a small study involving 10 subjects by Wilson et al. (1998), better comfort was reported for patients using randomly paired

lenses from Group II (high water content but non-ionic) and Group IV (high water content and ionic) FDA contact lenses (Jones et al., 2013).

Maïssa et al. (2012) conducted a study to investigate the impact of silicone hydrogel contact lenses on the ocular surface. They compared circumlimbal conjunctival staining and comfort levels among wearers of ACUVUE OASYS hydrogel silicone lenses (knife edge design), AIR OPTIX, Biofinity (chisel edge rounded edge combination), PureVision (rounded edge design), and ACUVUE 2 hydrogel lenses (knife edge design). Their findings indicated that rounded edge design lenses produced minimal circumlimbal staining but lower comfort levels, whereas knife edge design lenses resulted in higher circumlimbal staining but greater wearer comfort. However, the observed conjunctival staining and comfort levels were attributed to lens design rather than focusing solely on the material effects of different silicone hydrogel compositions.

Similarly, Efron et al. (1986), as cited in Jones et al. (2013), compared comfort levels among contact lenses based on water content. They found that lenses with lower water content (38%) were more comfortable than those with higher water content. Notably, the study excluded potential confounding factors such as lens edge design or surface finish, as all lenses were cut to the same shape and sourced from the same manufacturer.

Additionally, Young et al. (1997) conducted a study assessing comfort to predict successful contact lens wear. They evaluated lenses with low (38%), medium (54%-58%), and high (69%-74%) water content. Their findings recommended lenses with lower water content for greater wearing comfort.

Research on the evaluation of contact lens-related dehydration during initial application is extensive, as understanding the hydrating properties of hydrogel lenses is crucial due to various clinical implications. Dehydration can lead to changes in lens fit, discomfort, reduced oxygen transmission, and increased corneal drying (Nichols et al., 2002). Andrasko et al. (1983) reported that hydrogel lenses can dehydrate by 7%-11% during the first 30 minutes of wear, with thicker lenses exhibiting lower dehydration rates compared to thinner ones. Additionally, lenses with high water content experience more significant water loss than those with low water content, even at the same thickness.

The rate of oxygen absorption in the cornea is influenced by oxygen transmission (Dk) and lens thickness (t), with thinner lenses allowing more oxygen to reach the cornea (Jones & Dumbleton, 2019). Ideally, hydrogel lenses should have high oxygen transmission and thin central thickness.

However, this combination is impractical as it tends to lead to rapid dehydration and significant corneal staining (Jones & Dumbleton, 2019).

Maintaining a healthy ocular surface is essential for comfortable contact lens wear and to avoid serious complications. However, many contact lens wearers, even without underlying conditions such as blepharitis or meibomian gland dysfunction, report higher rates of dryness (Chalmers, 2014). The stability of the tear film and ocular surface greatly influences the success of contact lens

While there is no specific classification for hydrogel silicone contact lens groups, various materials such as somofilcon A, comfilcon A, fanfilcon A, samfilcon A, hilafilcon B, and others are utilized in their manufacture. Numerous studies have investigated the effects of wearing different material contact lenses on wearers. For instance, Iskeleli et al. (2013) compared tear evaluation before and after three months of wearing hydrogel silicone contact lenses from two different generations: Focus-Night & Day<sup>TM</sup> hydrogel silicone lenses for Group 1 and Air Optix <sup>TM</sup> silicone lenses for Group II. Statistical analysis indicated no significant differences between the two groups in terms of tear break-up time (TBUT) and Schirmer test values.

Similarly, Uğurlu et al. (2019) examined tear quantity and quality before the initial use of contact lenses and after one month and three months of wear. They compared Bausch & Lomb Ultra (samfilcon A) hydrogel silicone lenses on the right eye with Johnson-Johnson Vision Acuvue Oasys hydrogel silicone lenses (senofilcon A) on the left eye. No significant differences were observed in TBUT and Schirmer test values between the application of hydrogel silicone lenses made from samfilcon A and senofilcon A materials.

Date: 2/4/2024

#### 2.2 Problem statement and study justification

Since 2019, there has been limited research conducted in Malaysia regarding tear quality, corneal effects, and comfort levels associated with FDA contact lens groups. Recent studies in the realm of soft contact lenses have predominantly focused on silicone hydrogel varieties.

Existing literature indicates that contact lens application can alter tear layer parameters, although quantitative data on tear production resulting from contact lens wear has received scant attention (Downie & Craig, 2017; Razak et al., 2018). Information regarding tear quantity following 8 hours of contact lens wear is particularly lacking, necessitating further investigation into the effects of different contact lens types over longer durations (Razak et al., 2018).

Various contact lens brands exhibit differences in water content and thickness, with hydrogel lenses typically thinner than soft lenses with higher water content (Jones & Dumbleton, 2019). Notably, individuals may respond differently to lens thickness and water content variations. While some wearers may prefer thin lenses with low water content, others may find thicker lenses with medium or high water content more comfortable (Jones et al., 2013).

Since 2019, there has been limited research conducted in Malaysia regarding tear quality, corneal effects, and comfort levels associated with FDA contact lens groups. Recent studies in the realm of soft contact lenses have predominantly focused on silicone hydrogel varieties.

Existing literature indicates that contact lens application can alter tear layer parameters, although quantitative data on tear production resulting from contact lens wear has received scant attention (Downie & Craig, 2017; Razak et al., 2018). Information regarding tear quantity following 8 hours of contact lens wear is particularly lacking, necessitating further investigation into the effects of different contact lens types over longer durations (Razak et al., 2018).

Various contact lens brands exhibit differences in water content and thickness, with hydrogel lenses typically thinner than soft lenses with higher water content (Jones & Dumbleton, 2019). Notably, individuals may respond differently to lens thickness and water content variations. While some wearers may prefer thin lenses with low water content, others may find thicker lenses with medium or high water content more comfortable (Jones et al., 2013).

Differences in water content within soft contact lenses may contribute to corneal dehydration, leading to dryness in the eyes. Despite advancements in soft contact lens manufacturing, instances of corneal allergies or sensitivities to such lenses have been reported (Moreddu et al., 2019). Studies suggest that changes in the tear film may occur within the first hour of contact lens wear, but quantitative data on tear film thickness post-application is lacking (Nichols et al., 2004).

Furthermore, there is limited data available for tear assessment, corneal staining, and comfort levels among FDA contact lens groups I, II, III, and IV, with recent studies predominantly focusing on silicone hydrogel lenses. Therefore, this study aims to compare tear quality and quantity, as well as comfort levels, between these contact lens groups and silicone hydrogel lenses.

While tear assessment before and after wearing silicone hydrogel lenses may reveal significant changes, no substantial differences are observed between different silicone hydrogel materials. However, factors such as water content, material composition, wearing duration, and lens deposition are more closely associated with corneal staining than contact lens care solutions, ocular surface characteristics, tear composition, demographics, or medical factors (Nichols & Sinnott, 2011).

In response to consumer needs, advancements in contact lens technology continue, with efforts aimed at enhancing wearer comfort. Innovations such as the incorporation of wetting agents, hydrophilic monomers, surface treatments, and water gradient surface technology are introduced to mitigate the impact of wearing silicone hydrogel lenses on the tear layer (Sulley & Dumbleton, 2020). Therefore, ongoing research into technological and material developments in contact lens manufacturing is essential to understand their effects on consumers and to facilitate future improvements.

Date: 2/4/2024

#### 2.3 Research Questions

Is there a discrepancy in tear assessment, corneal staining, and comfort levels before and after one day (8 hours) of wearing FDA contact lenses Group I, II, III, IV, and V among undergraduate students at UKM Kuala Lumpur Campus?

#### 2.4 Research Hypothesis

Among UKM undergraduate students at the Kuala Lumpur Campus, there was no significant disparity observed in tear assessment, corneal staining, and comfort levels before and after one day (8 hours) of wearing Group I, II, III, IV, and silicone hydrogel contact lenses.

#### 2.5 Conceptual framework

Figure 1 illustrates the conceptual framework for assessing tear quantity, corneal staining, and comfort levels during the wear of FDA contact lenses Group I, II, III, IV, and V materials.



Date: 2/4/2024

## 2.6 Objectives

# 2.6.1 General Objectives:

The objective is to examine the impact of FDA contact lenses Group I, II, III, IV, and silicone hydrogel on tear assessment, corneal staining, and comfort levels among undergraduate students at UKM Kuala Lumpur Campus.

# 2.6.2 Specific Objectives:

i. Assessing tear quantity, corneal staining, and comfort levels before and after 8 hours of wearing FDA contact lenses Group I, II, III, IV, and silicone hydrogel.

ii. Contrasting tear evaluation and corneal staining pre- and post-8-hour application of FDA contact lenses Group I, II, III, IV, and silicone hydrogel.

iii. Comparing comfort levels pre- and post-8-hour wear among FDA contact lenses Group I, II, III, IV, and silicone hydrogel (Va and Vb).

#### 3.0 METHODOLOGISTS

#### 3.1.1 Study Design

The studies is a mixed, clinical trials and cross-sectional studies.

#### 3.1.2 Sampling Method

Random sampling is used in this study.

#### 3.1.3 Study Location

The study will take place at the Optometry Clinic within the Optometry and Vision Sciences Programme, Faculty of Health Sciences, Universiti Kebangsaan Malaysia. This location was selected due to its status as the primary clinic for optometry practice within the Faculty of Health Sciences, equipped with all necessary equipment for the study. Situated centrally within the Faculty of Health Sciences, it offers convenient access for undergraduate subjects participating in the study.

Date: 2/4/2024

# 3.1.4 Study Sample Calculation

The sample size for this study was determined using the Daniel formula (1999), with a total of 10% of the overall sample size allocated for the study. Considering a dropout rate of 10%, a total of 18 subjects were required for the study.

$$n = \frac{Z^2 P(1-P)}{d^2}$$

$$n = \frac{(1.96) (0.3)(1-0.3)}{(0.05)^{2}}$$

$$n = \frac{0.4116}{0.0025}$$

$$n = 164.64$$

n study = 
$$10\% \times 164.64$$

$$= 16.46$$

$$= 16$$

Dropout rate =  $10\% \times 16$ 

$$= 1.6$$

$$= 2$$

Total subjects = 16 + 2

= 18 subjects

n = required sample size

= 1.96, the value of Z when the confidence level is 95%  $Z^2$ 

P = 0.3, prevalence of contact lens clinic patients at UKM Optometry Clinic in semester 2, session 2022/2023

d = 0.05, margin of error

Date: 2/4/2024

### 3.1.5 Subject

UKM undergraduate students' Kuala Lumpur Campus was chosen as the subject of study because the location of the study was at the UKM Optometry Clinic located at the Kuala Lumpur Campus of UKM.

#### 3.1.6 Participation Criteria

- 1. Healthy volunteered individuals between 19 and 29 years old.
- 2. Individuals with a refraction power of less than -6.00 spherical diopters and astigmatism power of less than -1.00 cylindrical diopters.
- 3. Experienced contact lens wearers. (Participants are asked to lay off contact lenses for at least 2 weeks before the clinical trial starts (McKernan et al., 2014))

#### 3.1.7 Exclusion Criteria

- 1. Individuals who smoke (Ward et al. 2010)
- 2. Individuals with history of diseases on the ocular surface, ocular trauma, refractive surgery, intraocular and extraocular surgery.
- 3. Pregnant individuals (Yenerel &; Kucumen, 2015).
- 4. Individuals taking systemic drugs that can cause dry eyes (Fraunfelder et al. 2012).

#### 3.1.8 Instruments

- 1. Hydrogel soft contact lenses Group I, II, III, IV, Va and Vb
- 2. Schirmer Strip
- 3. Fluoresine Strip
- 4. Saline solution
- 5. Multipurpose solution Maxvue
- 6. Slitlamp Biomicroscope
- 7. Bausch & Lomb Keratometer
- 8. Contact Lens Discomfort Index Questionnaires (CLDI)

Date: 2/4/2024

3.1.9 Study Protocol

Participants for this study will be recruited from among UKM undergraduate students at the Kuala

Lumpur Campus based on the inclusion and exclusion criteria. Recruitment of volunteers will be

conducted through advertisement. Simple random sampling will be used for participant selection,

with those meeting the inclusion criteria being eligible for the study, while those meeting the

exclusion criteria will be dismissed.

Before the commencement of the clinical trial, all participants will be provided with a consent

form to review. The study will take place at the UKM Optometry Clinic, Jalan Raja Muda Abdul

Aziz, Kuala Lumpur, Malaysia.

Participants will be required to attend the UKM Optometry Clinic for three sessions, each lasting

8 hours, during which they will wear FDA hydrogel contact lenses (groups I, II, III, IV, Va and

Vb). Each lens will be placed on one eve only. Hence, the study will involve three wearing

sessions, with the first session focusing on groups I and II FDA contact lenses, the second session

on groups III and IV FDA contact lenses, and the third session on hydrogel silicone contact lenses

Va and Vb. A 2-week rest period will be provided between each session.

The complete study procedure is outlined as follows:

Care for Contact Lenses Leaflet.

Ensuring proper hygiene and technique is crucial to prevent eye health complications while

wearing contact lenses. Subjects will receive thorough guidance on essential practices, including:

maintaining hygiene care, correctly utilizing contact lens solution, applying and removing contact

lenses, and adhering to permissible actions during wear. Additionally, subjects will be provided

with a hotline for any inquiries or emergencies arising during contact lens use. Furthermore, they

will receive a pamphlet titled "Soft Contact Lens Instructions" available at the UKM KL

Optometry Clinic.

16



Figure 1 & 2. Soft contact lens use instructions

#### **Pre-Assessment**

A pre-assessment will precede the contact lens application during the initial session. The parameters measured will include these three tests: a) assessment of tear quantity using the Schirmer Test, b) evaluation of tear quality with the NIBUT Test, and c) examination of corneal staining using the Efron Grading Scale. These same tests will be conducted after the contact lenses have been worn for 8 hours and subsequently removed.

#### a) Tear Quantity Assessment (Schirmer Test)

To assess tear quantity, the Schirmer test will be employed using a 5mm x 30mm Schirmer strip. The strip will be positioned in the temporal area of the subject's lower eyelid. The subject will be instructed to look upwards and blink naturally for 5 minutes, after which the Schirmer strip will be removed. The length of the wet portion of the strip will be measured and documented. Three readings will be obtained in millimeters (mm), and the average reading will be calculated for data analysis (Kallarackal et al., 2002).

#### b) Tear Quality Assessment (NIBUT Test)

The assessment of tear quality was conducted using the Non-Invasive Break Up Time Test (NIBUT) technique with the Bausch & Lomb keratometer. The subject was instructed to rest their

chin on the designated chin rest and align their forehead with the headrest. Initially, the subject blinked several times and then refrained from blinking. Time was measured from the last blink until the appearance of any distortion or break in the "mires." This time interval was recorded as the NIBUT measurement. If the subject blinked during the measurement, the test was paused briefly, and resumed after a few blinks. A one to two-minute break was provided between each measurement. Three readings were taken, and the average of these readings was utilized for subsequent statistical analysis (Mohidin et al., 2002).

#### c) Corneal Coloring Assessment (Efron Grading Scale)

The evaluation of corneal staining will involve using the Efron Grading Scale to assess any marks or damage on the subject's cornea before applying contact lenses. Initially, fluorescein dye will be applied to the subject's eyes using fluorescein strips moistened with saline solution. The subject will be instructed to look up, and the moistened fluorescein strip will be gently touched to the lower eyelid, followed by blinking. Using a biomicroscopic slit lamp equipped with a blue cobalt light, any staining or markings on the cornea will be examined. Any observed findings will be documented according to the Efron Grading Scale. Subsequently, the subject's eyes will be rinsed with saline solution to remove the fluorescein dye. The cornea will be divided into five zones (central, superior, inferior, temporal, and nasal) for recording observations, as depicted in Figure 1. The Efron Grading Scale, recognized for its suitability in assessing corneal coloring, will guide the evaluation process (Dundas et al., 2001; Woods & Fonn, 2018). (Dundas et al., 2001; Woods & Fonn, 2018).



Date: 2/4/2024

Figure 3. Grading Scale Based on 5 Corneal Zones

# i. Contact lens application

The placement of group I FDA contact lenses will occur on one side of the subject's eye, while group II FDA contact lenses will be positioned on the opposite side, with the positioning being randomized and unknown to the subjects. Researchers will delicately insert the contact lenses, providing clear instructions and precautions to the subjects regarding their wear. Subjects will be advised to remain near the UKM KL Campus throughout the contact lens application and return to the UKM Optometry Clinic after 8 hours for lens removal. Additionally, subjects will be instructed to promptly notify the researcher of any discomfort, pain, or unforeseen issues related to the wearing of contact lenses.

#### ii. Post-Wear Assessment

The researcher will remove the contact lenses from the subject's eyes. Subsequently, a post-wearing examination of the contact lenses will be conducted. This examination mirrors the pre-use assessment and includes a) evaluating tear quantity using the Schirmer Test, b) assessing tear quality with the NIBUT Test, and c) grading corneal staining based on the Efron Grading Scale. Following the removal of contact lenses, subjects will be required to complete the Contact Lens Discomfort Index (CLDI) questionnaire twice at each appointment: once for the right eye and once for the left eye. This allows for the measurement of comfort levels separately for each eye.

#### d) Contact Lens Discomfort Index Questionaires (CLDI)

The CLDI questionnaire will be employed to evaluate the comfort level during the usage of Group I and II FDA contact lenses. This questionnaire's selection of questions is rooted in the Contact Lens Dry Eyes Questionnaire (CLDEQ)-8. Known for its robustness and reliability, the CLDI questionnaire is specifically crafted to gauge comfort levels associated with contact lens wear (Arroyo-del Arroyo et al., 2022).



Figure 4. Contact Lens Discomfort Index (CLDI) Questionnaire

#### i. Rest Period

A "washout period," also known as a rest period, lasting for two weeks will be provided to the subjects to prevent any unauthorized observations.

# ii. Second and Third Appointments

Subjects will be required to attend a second appointment following a rest period for the application of group III and IV FDA contact lenses. This appointment will involve the repetition of the procedure, including pre-application examination, contact lens wear, post-use examination, and subsequent rest period. The same procedure will be replicated for a third appointment involving the wearing of silicone hydrogel contact lenses Va and Vb.

#### 3.1.10 Flow Chart





#### 3.1.11 Data Analysis

The forthcoming study will employ IBM SPSS Statistics Version 27 for data analysis. The normality of the data will be assessed utilizing the Shapiro-Wilk test. Subsequently, the distribution of the data will be examined accordingly.

- i. Utilize the Paired t-test for normally distributed data or the Wilcoxon signed-rank test for non-normally distributed data to assess the disparities in tear quality and quantity before and after
- ii. Employ the Paired t-test for normally distributed data or the Wilcoxon signed-rank test for non-normally distributed data to compare the mean quality and quantity of tears between FDA contact lens application groups I and II, groups III and IV, as well as silicone hydrogel materials A and B.

Date: 2/4/2024

iii. Employ the Paired t-test for normally distributed data or the Wilcoxon signed-rank test

for non-normally distributed data to assess the comfort levels associated with the application of

FDA contact lenses within groups I and II, groups III and IV, as well as silicone hydrogel

materials A and B.

4.0 ETHICAL APPROVAL

Ethical approval has been approved by the UKM Research Ethics Committee, The National

University of Malaysia JEP-2023 679 (18 Dec 2023 – 18 March 2025).

24

Date: 2/4/2024

# **5.0 GANTT CHART**

| Year Activity (Month) | 2024 | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | JAN | FEB | MAR | APR | MAY | JUN | JUL | AUG | SEP | OCT | NOV | DEC |
| <b>Proposal Submission</b> | | | | | | | | | | | | |
| <b>Ethics Approval</b> | | | | | | | | | | | | |
| <b>Material Preparation</b> | | | | | | | | | | | | |
| Clinical Trial | | | | | | | | | | | | |
| Data Analysis | | | | | | | | | | | | |
| Manuscript Writing | | | | | | | | | | | | |
| Presentation | | | | | | | | | | | | |
| Manuscript | | | | | | | | | | | | |
| Submission | | | | | | | | | | | | |

#### 6.0 REFERENCES

 Arroyo, C. A., Fernández, I., La Rosa, A., Pinto-Fraga, J., González-García, M. J., & LópezMiguel, A. (2022). Design of a questionnaire for detecting contact lens discomfort: the Contact Lens Discomfort Index. Clinical and Experimental Optometry, 105(3), 268–274.

- 2. Asharlous, A., Jafarzadehpour, E., Mirzajani, A., Khabazkhoob, M., Heydarian, S. & Taghipour, A. 2016. Tear Deformation Time and optical quality in eyes wearing siliconee hydrogel contact lenses. Journal of Current Ophthalmology 28
- 3. Brautaset, R., Nilsson, M., Leach, N. E., Miller, W. R., Gire, A. I., Quintero, S., & Bergmanson, J. P. (2008). Corneal and Conjunctival Epithelial Staining in Hydrogel Contact Lens Wearers. Eye & Contact Lens-science and Clinical Practice, 34(6), 312–316.
- 4. Chalmers, R. L. (2014). Overview of factors that affect comfort with modern soft contact lenses. Contact Lens and Anterior Eye, 37(2), 65–76.
- Chatterjee, S. K., Upadhyay, P., Mishra, M., M, S., Akshara, M., Kamali, N., Zaidi, Z. S., Iqbal, S. F., & Misra, S. K. (2020). Advances in chemistry and composition of soft materials for drug releasing contact lenses. RSC Advances, 10(60), 36751–36777.
- 6. Chen, Q., Wang, J., Shen, M., Cai, C., Li, J., Cui, L., Qu, J. & Lu, F. 2009. Lower volumes of tear menisci in contact lens wearers with dry eye symptoms. Investigative Ophthalmology and Visual Science 50(7): 3159–3163.
- 7. Cope, J. R., Collier, S. A., Nethercut, H., Jones, J. M., Yates, K., & Yoder, J. S. (2017).
- 8. Risk Behaviors for Contact Lens-Related Eye Infections Among Adults and Adolescents United States, 2016. MMWR. Morbidity and mortality weekly report, 66(32), 841–845.
- 9. Craig, J. P., & Downie, L. E. (2019). Tears and Contact Lenses. In Elsevier eBooks (pp. 97–116).
- 10. Downie, L.E. & Craig, J.P. 2017. Tear film evaluation and management in soft contact lens wear: a systematic approach. Clinical and Experimental Optometry 100(5): 438–458.
- 11. Efron, N., Morgan, P. B., Maldonado-Codina, C., & Brennan, N. A. (2010). Contact lenses: the search for superior oxygen permeability. In Elsevier eBooks (pp. 280–303).

12. Fonn, D. 2007. Targeting contact lens-induced dryness and discomfort: What properties will make lenses more comfortable. Optometry and Vision Science 84(4): 279–285.

- 13. Fraunfelder, F. T., Sciubba, J. J., & Mathers, W. D. (2012). The role of medications in causing dry eye. Journal of Ophthalmology, 2012, 1–8.
- 14. Gasson, A. & Morris, J. 2003. The Contact Lens Manual: A Practical Guide to Fitting. The Contact Lens Manual: A Practical Guide to Fitting. Butterworth-Heinemann.
- 15. Heiting, G., OD. (2019). What are contacts made of? All About Vision.
- 16. Iskeleli, G., Karakoc, Y., Ozkok, A., Arici, C., Ozcan, O. & Ipcioglu, O. 2013. Comparison of the effects of first and second generation silicone hydrogel contact lens wear on tear film osmolarity. International journal of Ophthalmology 6(5): 666–670.
- 17. Jones, L., & Dumbleton, K. (2019). Soft Contact Lens Fitting. In Elsevier eBooks (pp. 207–222).
- Jones, L., Brennan, N. A., González-Méijome, J. M., Lally, J., Maldonado-Codina, C., Schmidt, T. A., Subbaraman, L. N., Young, G. P., & Nichols, J. J. (2013). The TFOS International Workshop on Contact Lens Discomfort: Report of the Contact Lens Materials, Design, and Care Subcommittee. Investigative Ophthalmology & Visual Science, 54(11), TFOS37.
- 19. Kallarackal, G.U., Ansari, E.A., Amos, N., Martin, J.C., Lane, C. & Camilleri, J.P. 2002. A comparative study to assess the clinical use of Fluorescein Meniscus Time (FMT) with Tear Break up Time (TBUT) and Schirmer's tests (ST) in the diagnosis of dry eyes. Eye 16(5): 594–600.
- 20. Kim, E., Saha, M. & Ehrmann, K. 2018. Mechanical Properties of Contact Lens Materials. Eye & Contact Lens 44(July 2018): S148–S156.
- 21. Krejcie, R. V. & Morgan, D.W. 1970. Determining Sample Size for Research Activities. Educational and Psychological Measurement 30(3): 607–610.
- 22. Lakkis, C., & Brennan, N. A. (1996). Bulbar conjunctival fluorescein staining in hydrogel contact lens wearers. The CLAO journal: official publication of the Contact Lens Association of Ophthalmologists, Inc, 22(3), 189–194.
- 23. Lemp, M.A. 1995. Report of the National Eye Institute/Industry Workshop on Clinical Trials in Dry Eyes. CLAO Journal 21(4): 221–232.
- 24. Lloyd McKernan, A., O'Dwyer, V. & Simo Mannion, L. 2014. The influence of soft contact lens wear and two weeks cessation of lens wear on corneal curvature. Contact Lens and Anterior Eye 37(1): 31–37.

25. Maïssa, C., Guillon, M. & Garofalo, R.J. 2012. Contact lens-induced circumlimbal staining in siliconee hydrogel contact lenses worn on a daily wear basis. Eye & contact lens 38(1): 16–26.

- 26. Maruyama, K., Yokoi, N., Takamata, A. & Kinoshita, S. 2004. Effect of environmental conditions on tear dynamics in soft contact lens wearers. Investigative Ophthalmology and Visual Science 45(8): 2563–2568.
- 27. Mohidin, N., Bay, T.C. & Yap, M. 2002. Non-invasive tear break-up time in normal Malays. Clinical and Experimental Optometry 85(1): 37–41.
- 28. Moreddu, R., Vigolo, D., & Yetisen, A. K. (2019). Contact Lens Technology: From Fundamentals to Applications. Advanced Healthcare Materials, 8(15), 1900368.
- 29. Mutalib H. A., and Lim, Y. V. (2018) Ocular comfort assessment in hydrogel and siliconee hydrogel contact lens wearers. Jurnal Sains Kesihatan Malaysia, 16 (2). pp. 65-69. ISSN 1675-8161
- 30. Nichols, K. K., Mitchell, G. E., Simon, K. M. S., Chivers, D. A., & Edrington, T. B. (2002). Corneal Staining in Hydrogel Lens Wearers. Optometry and Vision Science, 79(1), 20–30.
- 31. Nichols, J. J., & King-Smith, P. E. (2004). The Impact of Hydrogel Lens Settling on the Thickness of the Tears and Contact Lens. Investigative Ophthalmology & Visual Science, 45(8), 2549.
- 32. Nichols, J. J., & Sinnott, L. T. (2006). Tear film, contact lens, and patient-related factors associated with contact lens-related dry eye. Investigative ophthalmology & visual science, 47(4), 1319–1328.
- 33. Nichols, J.J. & Sinnott, L.T. 2011. Tear film, contact lens, and patient fact